CLINICAL TRIAL: NCT01990066
Title: Single Institution Randomized Controlled Study of a Home Based Exercise Program to Reduce Functional Decline, Cancer Related Fatigue (CRF and Improve Quality of Life for the Elderly Gynecologic Oncology Patient)
Brief Title: Home Based Exercise Program for Elderly Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting adequate enrollment
Sponsor: Duke University (Other)
Collaborators: Oncology Nursing Centers for Excellence (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00046121
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-11

CONDITIONS: Cancer Related Fatigue
Keywords: Quality of Life; Physical Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Subjects randomized to intervention will receive Physical Therapist instructed exercise teaching. They will receive a home exercise DVD and flip ring of exercises. Subjects will be asked to perform home exercise 3 days weekly consisting of 13 strengthening/stretching exercises and 20 mins of aerobic exercise, walking or seated aerobics using ergometer. Subjects will record their exercise on a log and return on day 1 of every cycle.
  Interventions: Behavioral: Home Based Exercise
- Observation (No Intervention): Subjects randomized to observation will only have physical therapy assessment using the Berg Balance Test and 6min Walk Test at baseline and end point. These subjects will not receive any exercise teaching.

INTERVENTIONS:
Behavioral: Home Based Exercise — Subjects randomized to intervention will receive Physical Therapist instructed exercise teaching. They will receive a home exercise DVD and flip ring of exercises. Subjects will be asked to perform home exercise 3 days weekly consisting of 13 strengthening/stretching exercises and 20 mins of aerobic exercise, walking or seated aerobics using ergometer. Subjects will record their exercise on a log and return on day 1 of every cycle.
  Arms: Intervention

SUMMARY:
Implementation of a home based exercise program to reduce functional decline, cancer related fatigue (CRF) and improve quality of life in the elderly gynecologic oncology patient

Problem:

Can prevention of CRF and loss of function improve QOL in the elderly gynecologic oncology patient undergoing chemotherapy?

Support:

Fatigue and its impact on QOL is a major concern with the elderly patient receiving chemotherapy. When compared to younger adults QOL is more important than gain in survival for elderly patients. (Eyigor, et al., 2010).

The National Comprehensive Cancer Network recommends exercise as the most effective intervention for cancer related fatigue.

Methods:

This is a single institution randomized controlled study to evaluate a home based exercise program in elderly gynecologic oncology patients undergoing chemotherapy. Subjects will be randomized to the intervention group or to the control group receiving usual care.

Intervention group will receive a home exercise program 3 days weekly consisting of 30mins of strength and aerobic activity, utilizing a follow along exercise DVD and patient log to assist with compliance.

The two groups will be compared by 1) objective PT assessment with the Berg Balance and 6 minute walk test (before or after) Cycle 1 and 6, 2) subjective nursing assessment with the NHANES (National Health and Nutrition Examination Survey) and FACIT- F (Functional Assessment of Chronic Illness Therapy: Fatigue) prior to Cycle 1 (baseline),4 (midpoint), and following cycle 6 (completion).

Conclusion:

PT directed home exercise program may improve CRF, functional decline, and QOL in elderly gynecologic oncology patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial, Ovarian, Cervix, Vaginal Cancer Initiating Chemotherapy
* Age greater than or equal to 65yrs
* ECOG (Eastern Cooperative Oncology Group) performance status less than 3
* No current physical therapy intervention
* English speaking

Exclusion Criteria:

* Non-gynecologic malignancy
* Recurrent cancer
* Receiving radiation alone
* Gait or balance disturbance

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduction in Cancer Related Fatigue (CRF) | Baseline, +/- 7days of 4th chemo cycle (mid point), +/- 7 days of 3 weeks after 6th cycle (end point)
  CRF will be evaluated using the FACIT-F tool.

SECONDARY OUTCOMES:
Quality of Life Improvement (QOL) | Baseline, +/- 7days of cycle 4 of treatment (mid point), +/- 7 days of 3rd week after cycle 6 (end point)
  QOL will be evaluated using the NHANES and FACIT-F tools.
Reduction in Physical Functional Decline | Baseline and +/- 7days of 3 weeks post 6th cycle (end point)
  Physical function will be evaluated using the Berg Balance Test and 6 Min Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Alicia S. Johnson, ADN-RN, Principal Investigator — Duke University
Locations (1):
- Duke Raleigh Cancer Center, Raleigh, North Carolina, United States